CLINICAL TRIAL: NCT00706550
Title: Immune Responses to Pneumococcal Vaccination Among HIV-Infected Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Albert Einstein College of Medicine (Other); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INDA-002-08S
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Results first posted 2013-12-12 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infections
Keywords: pneumococcal polysaccharide vaccine
MeSH Terms: conditions — HIV Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate (Other): Arm 1 will receive PV (23-valent pneumococcal polysaccharide vaccine) prior to starting antiretroviral treatment and will receive PLACEBO after at least 6 months of starting antiretroviral treatment.
  PV (23-valent pneumococcal polysaccharide vaccine): Currently commercially available pneumococcal polysaccharide vaccine
  Interventions: Biological: (PV) 23-valent pneumococcal polysaccharide vaccine; Biological: Placebo
- Delayed (Other): Arm 2 will receive PLACEBO prior to starting antiretroviral treatment and will receive PV (23-valent pneumococcal polysaccharide vaccine) after at least 6 months of starting antiretroviral treatment.
  PV (23-valent pneumococcal polysaccharide vaccine): Currently commercially available pneumococcal polysaccharide vaccine
  Interventions: Biological: (PV) 23-valent pneumococcal polysaccharide vaccine; Biological: Placebo

INTERVENTIONS:
Biological: (PV) 23-valent pneumococcal polysaccharide vaccine — Currently commercially available pneumococcal polysaccharide vaccine
  Other Names: Pneumovax 23
Biological: Placebo — Placebo

SUMMARY:
The purpose of this study is to evaluate the best timing for administering pneumococcal vaccine (PV) to HIV-infected adults that have CD4 cell counts of more than 200 and are not yet receiving combination antiretroviral treatment (ART). Participants in this study will be assigned by chance to receive vaccination with PV prior to starting ART or after at least 6 months of ART. Antibody levels to components of the PV will be measured at 6 months and 12 months after vaccination. The results will tell us if patients that receive PV after 6 months of ART have better response to the vaccine than those that get vaccinated prior to treatment.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count >200
* no acute illness
* no pneumococcal vaccination within 3 years
* naive to treatment or if previously on treatment, no antiretroviral treatment for at least 6 months
* willingness to start antiretroviral treatment as recommended by current guidelines

Exclusion Criteria:

* prior pneumococcal vaccination within 3 years
* prior AIDS diagnosis based on opportunistic disease
* acute illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Rodriguez-Barradas, MD, Principal Investigator — Michael E. DeBakey VA Medical Center
Locations (1):
- Michael E DeBakey VA Medical Center, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 107 patients were enrolled on the study (11/2008-2/2011 at the Michael E. DeBakey VA Medical Center, at Thomas Street Clinic and at Legacy Clinic, in Houston, TX. Only the patients that completed the 1 month post-PV visit are included in the analysis (N=36 for each arm for a total of 72 out of the 107 initially enrolled).
Groups:
- Immediate: PV Before Starting Antiretroviral Therapy: Immediate group (Arm 1) received PV prior to starting antiretroviral treatment.
  PV (23-valent pneumococcal polysaccharide vaccine): Currently commercially available pneumococcal polysaccharide vaccine.
- Delayed: PV After >6 Months of Antiretroviral Therapy: Delayed group (Arm 2) received PV after at least 6 months of antiretroviral treatment
  PV (23-valent pneumococcal polysaccharide vaccine): Currently commercially available pneumococcal polysaccharide vaccine.
Period: Overall Study
Arm/Group | Immediate: PV Before Starting Antiretroviral Therapy | Delayed: PV After >6 Months of Antiretroviral Therapy
Started | 43 | 64
Completed | 36 | 36
Not Completed | 7 | 28

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: PV Before Starting Antiretroviral Therapy: Arm 1 received PV prior to starting antiretroviral treatment.
  PV (23-valent pneumococcal polysaccharide vaccine): Currently commercially available pneumococcal polysaccharide vaccine
- Arm 2: PV After >6 Months of Antiretroviral Therapy: Arm 2 received PV after at least 6 months of antiretroviral treatment.
  PV (23-valent pneumococcal polysaccharide vaccine): Currently commercially available pneumococcal polysaccharide vaccine
- Total: Total of all reporting groups
Arm/Group | Arm 1: PV Before Starting Antiretroviral Therapy | Arm 2: PV After >6 Months of Antiretroviral Therapy | Total
Number analyzed (Participants) | 43 | 64 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 63 | 105
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (12.9) | 40.8 (11.6) | 41.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 21
  Male | 37 | 49 | 86
Region of Enrollment [Number; unit: participants]
  United States | 43 | 64 | 107

OUTCOME MEASURES:

1. Primary Outcome: Immunoglobulin G (IgG) Levels
Description: Immunoglobulins are antibodies or special proteins that the immune system produces to protect the body against infections. IgG is the most common antibody. We measure baseline levels (before the vaccine is administered) to know how much antibody the subject has at the start point to be able to evaluate how much antibody is produced after the vaccine is administered.
Time Frame: Baseline
Measure: Geometric Mean (Full Range); unit: Micrograms/ml
Arm/Group | Immediate: PV Before Starting Antiretroviral Therapy | Delayed: PV After >6 Months of Antiretroviral Therapy
Number analyzed (Participants) | 36 | 36
Micrograms/ml
  IgG levels against CPS 6B | 5.12 (1.0) [0.71 to 27.60] | 5.17 (1.0) [1.10 to 22.87]
  IgG levels against CPS 23F | 1.80 (1.0) [0.44 to 9.35] | 1.83 (1.0) [0.74 to 4.71]

2. Primary Outcome: IgG Levels
Description: Immunoglobulins are antibodies or special proteins that the immune system produces to protect the body against infections. IgG is the most common antibody. This point of time (one-month after vaccine), gives the information about how much antibody was produced by the participant's immune system in response to the vaccine.
Time Frame: One-month post-vaccine
Measure: Geometric Mean (Full Range); unit: Micrograms/ml
Arm/Group | Immediate: PV Before Starting Antiretroviral Therapy | Delayed: PV After >6 Months of Antiretroviral Therapy
Number analyzed (Participants) | 36 | 36
Micrograms/ml
  IgG levels against CPS 6B | 7.85 (1.0) [2.94 to 43.58] | 5.79 (1.0) [1.23 to 21.42]
  IgG levels against CPS 23F | 2.50 (1.0) [0.62 to 23.37] | 2.41 (1.0) [0.80 to 7.94]

3. Primary Outcome: Immunoglobulin M (IgM) Levels
Description: Immunoglobulins are antibodies or special proteins that the immune system produces to protect the body against infections. IgM is the first antibody produced by the immune system to fight a new infection. We measure baseline levels (before the vaccine is administered) to know how much antibody the subject has at the start point to be able to evaluate how much antibody is produced after the vaccine is administered.
Time Frame: Baseline
Measure: Geometric Mean (Full Range); unit: Micrograms/ml
Arm/Group | Immediate: PV Before Starting Antiretroviral Therapy | Delayed: PV After >6 Months of Antiretroviral Therapy
Number analyzed (Participants) | 36 | 36
Micrograms/ml
  IgM levels against CPS 6B | 1.89 [0.40 to 7.56] | 1.85 [0.39 to 4.86]
  IgM levels against CPS 23F | 0.59 [0.01 to 4.29] | 0.78 [0.09 to 3.18]

4. Primary Outcome: IgM Levels
Description: Immunoglobulins are antibodies or special proteins that the immune system produces to protect the body against infections. IgM is the first antibody produced by the immune system to fight a new infection. This point of time (one-month after vaccine), gives the information about how much antibody was produced by the participant's immune system in response to the vaccine.
Time Frame: One-month post-vaccine
Measure: Geometric Mean (Full Range); unit: Micrograms/ml
Arm/Group | Immediate: PV Before Starting Antiretroviral Therapy | Delayed: PV After >6 Months of Antiretroviral Therapy
Number analyzed (Participants) | 36 | 36
Micrograms/ml
  IgM levels against CPS 6B | 2.18 [0.42 to 9.00] | 2.26 [0.59 to 6.29]
  IgM levels against CPS 23F | 0.65 [0.02 to 3.20] | 0.84 [0.23 to 2.86]

5. Primary Outcome: Opsonophagocytic Killing Activity (OPA)
Description: This assay helps us to know how the antibody produced by the body are working to kill the bacteria against which the antibody is produced. As explained previously for the immunoglobulins' assays, we measure the baseline point to be able to determine the increase after the vaccine is administered.
Time Frame: Baseline
Measure: Geometric Mean (Full Range); unit: Titers
Arm/Group | Immediate: PV Before Starting Antiretroviral Therapy | Delayed: PV After >6 Months of Antiretroviral Therapy
Number analyzed (Participants) | 23 | 36
Titers
  OPA titers against CPS 6B | 4.5 [2 to 512] | 6.0 [2 to 512]
  OPA titers against CPS 23F | 2.9 [2 to 32] | 2.9 [2 to 256]

6. Primary Outcome: Opsonophagocytic Killing Activity (OPA)
Description: This assay helps us to know how the antibody produced by the body are working to kill the bacteria against which the antibody is produced. This point of time (one-month after vaccine), gives the information about how much the killing activity increased 1 month after the vaccine was administered.
Time Frame: One-month post-vaccine
Measure: Geometric Mean (Full Range); unit: Titers
Arm/Group | Immediate: PV Before Starting Antiretroviral Therapy | Delayed: PV After >6 Months of Antiretroviral Therapy
Number analyzed (Participants) | 23 | 36
Titers
  OPA titers against CPS 6B | 23.0 [2 to 512] | 13.7 [2 to 512]
  OPA titers against CPS 23F | 4.7 [2 to 128] | 3.3 [2 to 64]

ADVERSE EVENTS:
Arm/Group | Arm 1: PV Before Starting Antiretroviral Therapy | Arm 2: PV After >6 Months of Antiretroviral Therapy
Serious Adverse Events (participants affected / at risk) | 6/43 | 8/64
Other Adverse Events (participants affected / at risk) | 2/43 | 1/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: PV Before Starting Antiretroviral Therapy (N=43) | Arm 2: PV After >6 Months of Antiretroviral Therapy (N=64)
CHF, arrhythmia (Cardiac disorders) | 1 (1) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 2 (2)
Dehydration, electrolite abnormalities (General disorders) | 0 (0) | 1 (2)
Elective surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Gastrointestinal infections and other disorders (Gastrointestinal disorders) | 0 (0) | 2 (5)
Mental health related (Psychiatric disorders) | 2 (3) | 0 (0)
Other infections (Infections and infestations) | 1 (1) | 1 (2)
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1: PV Before Starting Antiretroviral Therapy (N=43) | Arm 2: PV After >6 Months of Antiretroviral Therapy (N=64)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes